CLINICAL TRIAL: NCT03009279
Title: Relationship of Metabolic Syndrome and Its Components With Thyroid Nodule(s)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lin Liao (Other)
Responsible Party: Sponsor-Investigator, Lin Liao, chief of endocrinology department at Qianfoshan Hospital, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: qfsnfm-004
Record Dates: First submitted 2016-12-26; First posted 2017-01-04 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Metabolic Syndrome; Thyroid Nodule
Keywords: blood pressure; fasting plasma glucose; thyroid stimulating hormone
MeSH Terms: conditions — Metabolic Syndrome; Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- The MS group: Patients with metabolic syndrome(MS).
- The non-MS group: Patients without metabolic syndrome(MS).

SUMMARY:
To investigate the association between metabolic syndrome (MS) and thyroid nodule(s).

DETAILED DESCRIPTION:
To investigate the association between metabolic syndrome (MS), body mass index (BMI), hyperglycemia, dyslipidemia, hypertension and thyroid nodule(s) or thyroid functions in euthyroid subjects. Screen for the risk factors that affect the incidence of thyroid nodule(s).

ELIGIBILITY:
Inclusion Criteria:

1. People who received routain physical and laboratory examinations in the Health Management Cenre of QianFoShan Hospital from Jan. 2013 to Dec. 2015.
2. signed the informed consent.
3. Have complete clinical data.

Exclusion Criteria:

1. Patients with previous history of thyroid disease other than thyroid nodules.
2. People with abnormal thyroid function.
3. Thyroid ultrasound revealed patients with other lesions other than normal thyroid and thyroid nodules.
4. Pregnant or lactating women.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People who received routain physical and laboratory examinations in the Health Management Cenre of QianFoShan Hospital from Jan. 2013 to Dec. 2015.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The laboratory examinations | In 2013-2015
  Lipids,glucose,thyroid functions

SECONDARY OUTCOMES:
Blood pressure of patients in each group | In 2013-2015

OTHER OUTCOMES:
BMI of patients in each group | In 2013-2015
  body mass index（BMI）
Age of patients in each group | In 2013-2015
Gender of patients in each group | In 2013-2015

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, Study Chair — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Yes